CLINICAL TRIAL: NCT01966926
Title: Self-Weighing Instruction Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0807S41483
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Weight Loss; Body Weight
Keywords: self monitoring; self weighing; weight tracking; psychosocial outcomes; feasibility
MeSH Terms: conditions — Weight Loss; Body Weight | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily Weight Tracking (Experimental): weighing frequency instructions and tips
  Interventions: Behavioral: weighing frequency instructions and tips
- Weekly Weight Tracking (Experimental): weighing frequency instructions and tips
  Interventions: Behavioral: weighing frequency instructions and tips

INTERVENTIONS:
Behavioral: weighing frequency instructions and tips — Weekly emails with nutrition, physical activity, and weight tracking tips sent for 24 weeks

SUMMARY:
Scant data have been reported on the effects of weight self-monitoring during weight control. The purpose of this pilot project was to consider the questions: Is it possible to assign participants to engage in daily weight self-monitoring, and are there differential effects on mood of daily versus weekly weighing?

DETAILED DESCRIPTION:
This study tested the feasibility of assigning participants to daily or weekly weighing, monitored adherence to weighing instructions, and tracked additional behavioral and psychosocial indicators over a period of six months. It was hypothesized that there would be no differences in mood or adherence between daily versus weekly weighing conditions. Knowledge about the benefits of frequent self-weighing may shape public health recommendations for regular weighing as a weight reduction or obesity prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 25 and 35 kg/m2

Exclusion Criteria:

* Current weight loss program participation
* Chronic health conditions (diabetes, cancer, heart disease, psychiatric disorders requiring medication)
* Current or past eating disorder
* Current pregnancy or pregnant in past year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Linde, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited in Sept-Oct 2009 from craigslist.com ads and flyers in a University of Minnesota office building. 58 contacted the study and 28 were excluded [did not complete screening (n=10), not eligible due to weight or health exclusions (n=15), or withdrew before consent (n=3)], resulting in a final sample of 30 participants.
Groups:
- Daily Weight Tracking: daily weighing frequency instructions and tips
- Weekly Weight Tracking: weekly weighing frequency instructions and tips
Period: Overall Study
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (9.5) | 46.4 (13.8) | 45.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) was calculated from height and weight measured by the investigator at baseline.
  kg/m^2 | 30.99 (2.97) | 31.08 (3.37) | 31.04 (3.12)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Weight Tracking Instructions
Description: Participants were assigned to daily or weekly weight tracking, and were asked to return postcards once a week with weights recorded (7 for daily, 1 for weekly).
Time Frame: 6 months
Population: All participants were included in the analysis.
Measure: Number; unit: percentage of postcards returned
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 15 | 15
percentage of postcards returned | 98.3 | 96.7
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = .15, Chi-squared — P-value was unadjusted, with an a priori threshold for statistical significance set at p <.05; 1 degree of freedom; chi square = 2.05

2. Secondary Outcome: Changes in Depression Ratings
Description: Ratings of depressed mood, assessed by the Beck Depression Inventory, were obtained at baseline, three, and six months; the comparison of depression scores between groups and over time from baseline to 3 and 6 months was considered as a secondary outcome and analyzed using repeated measures multivariate analysis of variance (MANOVA). Scores on the inventory range from 0 to 63, with higher scores indicating greater presence of depressive symptoms. Scores from 0-10 represent normal mood; 11-16 = mild mood disturbance; 17-20 = borderline clinical depression; 21-30 = moderate depression; 31-40 = severe depression; > 40 = extreme depression.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 15 | 15
units on a scale
  baseline depression | 3.6 (3.5) | 6.3 (4.4)
  3-month depression | 3.9 (4.4) | 7.1 (4.1)
  6-month depression | 4.8 (5.6) | 6.7 (6.1)
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Repeated measures analysis from baseline to six months; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = 0.61, MANOVA — P-value not adjusted for multiple comparisons; a priori threshold of <0.05 for statistical significance; Degrees of freedom: 2,27; Wilks' Lambda = 0.96

3. Secondary Outcome: Changes in Anxiety
Description: Ratings of anxiety, assessed by the Beck Anxiety Inventory, were assessed at baseline, three, and six months; a comparison of anxiety scores between groups and over time from baseline to 3 and 6 months was considered a secondary outcome and analyzed using repeated measures MANOVA. Possible scores on the scale range from 0-63. Scores from 0-7 indicate minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 15 | 15
units on a scale
  baseline anxiety | 2.3 (2.9) | 5.7 (5.0)
  3-month anxiety | 2.7 (3.5) | 5.8 (4.5)
  6-month anxiety | 3.9 (6.0) | 5.3 (4.6)
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Repeated measures analysis from baseline to six months; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = 0.50, MANOVA — P-value is unadjusted; a priori threshold for statistical significance was <0.05; Degrees of freedom: 2,27; Wilks' Lambda = 0.95

4. Secondary Outcome: Changes in Body Image
Description: Changes in self-reported body image were assessed at baseline, three, and six months using the Appearance subscale of the Multidimensional Body Image Questionnaire. The subscale has a range of 0 to 42, with higher scores indicating better body image. A comparison of body image scores between groups and over time from baseline to 3 and 6 months was considered a secondary outcome and analyzed using repeated measures MANOVA.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 15 | 15
units on a scale
  baseline body image | 20.1 (7.0) | 19.1 (8.0)
  3-month body image | 22.6 (4.9) | 17.9 (8.6)
  6-month body image | 21.4 (5.9) | 18.5 (8.7)
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Repeated measures analysis from baseline to six months; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = 0.15, MANOVA — P-value not adjusted for multiple comparisons; a priori threshold for statistical significance was <0.05; Degrees of freedom: 2,27; Wilks' Lambda = 0.87

5. Secondary Outcome: Changes in Barriers to Weight Tracking
Description: Perceived barriers to self-weighing were assessed at baseline, three, and six months using a scale created for this study. The scale has a range of 18 to 90, with higher scores indicating greater perceptions of barriers to self-weighing. A comparison of barriers scores between groups and over time from baseline to 3 and 6 months was considered a secondary outcome and analyzed using repeated measures MANOVA.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 14 | 15
units on a scale
  baseline barriers | 39.7 (13.1) | 46.7 (14.7)
  3-month barriers | 27.5 (9.0) | 37.3 (9.5)
  6-month barriers | 30.7 (12.9) | 34.3 (12.4)
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Repeated measures analysis from baseline to six months; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = 0.30, MANOVA — P-value not adjusted for multiple comparisons; a priori threshold for statistical significance was <0.05; Degrees of freedom: 2,26; Wilks' Lambda = 0.91

6. Secondary Outcome: Changes in Perceptions of Weight Tracking
Description: Perceptions of weight tracking (ease of remembering and understanding, usefulness, awareness, interest, reward value, satisfaction, motivational value) were assessed at three and six months using a scale created for the study. The scale has a range of 0 to 64, with higher scores indicating greater perceptions of favorability of weight tracking. A comparison of perceptions scores between groups and over time from 3 and 6 months was considered a secondary outcome and analyzed using repeated measures MANOVA.
Time Frame: three to six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Number analyzed (Participants) | 15 | 15
units on a scale
  3-month perceptions | 47.7 (10.6) | 40.4 (10.2)
  6-month perceptions | 48.2 (10.0) | 45.0 (7.7)
Statistical Analysis 1: Comparison: Daily Weight Tracking vs Weekly Weight Tracking; Repeated measures analysis from three to six months; Test type: Non-Inferiority or Equivalence — Power not calculated due to small sample size and pilot study intent; p = 0.17, MANOVA — P-value not adjusted for multiple comparisons; a priori threshold for statistical significance was <0.05; Degrees of freedom: 1,28; Wilks' Lambda = 0.93

ADVERSE EVENTS:
Arm/Group | Daily Weight Tracking | Weekly Weight Tracking
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size; Absence of instructions that would mimic a weight loss program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes